CLINICAL TRIAL: NCT04555590
Title: Implementation of an Evidence Based Parentally Administered Intervention for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Duke University (Other); University of Chicago (Other); Wake Forest University Health Sciences (Other); Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Rosemary White-Traut, Director of Nursing Research and Evidence Based Practice, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00035600; 1R01HD098095-01A1 (NIH)
Record Dates: First submitted 2020-08-19; First posted 2020-09-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Premature Infants; Parent-Child Relations
Keywords: Premature Infants; NICU; Parental Stress; Healthcare Costs
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: This is an implementation study of the H-HOPE Intervention. The team uses a Stepped-Wedge Design for Implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre H-HOPE Cohort (No Intervention): The Pre-H-HOPE Comparison Cohort will not receive the H-HOPE intervention, and represents the prior standard (non-HOPE).
- H-HOPE Cohort (Experimental): The H-HOPE Cohort will receive the H-HOPE intervention.
  Interventions: Behavioral: H-HOPE Intervention

INTERVENTIONS:
Behavioral: H-HOPE Intervention — The H-HOPE intervention (Hospital to Home: Optimizing the Preterm Infant's Environment) to promote early infant development and parental engagement. H-HOPE includes ATVV, which provides Auditory (voice), Tactile (moderate touch massage), Visual (eye to eye), and Vestibular (rocking) stimulation with a parent-directed component which provides participatory guidance and social support to engage with their infants.
  Arms: H-HOPE Cohort

SUMMARY:
Early developmentally-based behavioral intervention has well-established positive effects and is recommended as the standard of care to support early brain maturation, health, and development. However, few neonatal intensive care units (NICUs) provide this early intervention. H-HOPE (Hospital to Home: Optimizing the Preterm Infant's Environment) has established efficacy, and has a standardized protocol, making it ready for widespread implementation. The infant-directed component of H-HOPE provides Auditory (voice), Tactile (moderate touch massage), Visual (eye to eye), and Vestibular (rocking) stimulation starting when infants are ready for social interaction. The parent-directed component of H-HOPE includes participatory guidance and support to help parents engage with infants in the NICU and the transition to home. In this NIH-funded research, H-HOPE improved growth, developmental maturity and mother-infant interaction, and reduced initial hospitalization costs and acute care visits through 6-weeks corrected age. This research tests whether H-HOPE can be implemented and sustained in five diverse NICUs, using a Type 3 Hybrid design to evaluate both implementation processes and effectiveness. The specific aims are to: 1) Identify the degree of implementation success; 2) Evaluate the effectiveness of H-HOPE for infants, hospital costs from H-HOPE enrollment until discharge, and parents, compared to a pre-implementation comparison cohort; and 3) Determine influences (facilitators and barriers) associated with implementation success and H-HOPE effectiveness, guided by the Consolidated Framework for Implementation Research (CFIR). An incomplete stepped-wedge design guides staggered roll-out for five clinical sites. Each NICU completes the CFIR implementation steps (Planning and Engaging, Executing, and Reflecting and Evaluating), followed by 6 months of Sustaining. For Aim 1, degree of implementation success is determined every two months as Sustainability (still offering H-HOPE), Reach (% of eligible parent/infant dyads receiving H-HOPE) and Degree of Implementation (mean H-HOPE services received per parent-infant unit) (primary implementation outcomes). For Aim 2, effectiveness is analyzed using generalized linear mixed models for infant, cost, and parent outcomes (primary outcomes: infant growth at discharge and acute care visits from discharge to 6-weeks corrected age). Propensity score analysis is used to make the pre- and post-implementation comparable. For Aim 3, a mixed methods analyses is used to identify influences from H-HOPE records and interviews that are associated with implementation success and effectiveness at each site and across sites. This is the first time implementation in a NICU is guided by the evidence-based CFIR framework, and results will make a major contribution to implementation science. This study will produce an evidence-based implementation strategy and Toolkit to disseminate nationwide. Widespread H-HOPE implementation will make a significant change in clinical practice and improve preterm infant health and health care costs.

ELIGIBILITY:
There are two cohorts of infants and parents: the Pre-H-HOPE Comparison Cohort and H-HOPE Cohort. H-HOPE is a family intervention, so parent(s) and infants are recruited together and must meet both parent and infant eligibility criteria. Infant and parent eligibility criteria are the same for both cohorts (Pre-H-HOPE and H-HOPE). Additionally, there are criteria for hospital personnel.

Inclusion criteria for the infant:

* born between 23-35 weeks gestational age (GA)
* have reached 31-32 weeks post menstrual age (PMA)
* clinically stable
* male or female
* could be receiving oxygen or intravenous therapy
* could have been previously intubated for mechanical ventilation
* assessed as ready to begin social interaction Infants of multiple births will be eligible to participate but data from only one randomly selected infant will be used in analysis of Aim 2.

Inclusion criteria for the parent (up to 2 per infant can be in the study:

* mother, father, other family member, or surrogate parent regardless of age, race/ethnicity, gender, or sexual orientation, or biological relationship to the infant
* intends to act in the role of parent
* 18 years of age or older
* English or Spanish speaking

Inclusion criteria for hospital personnel:

Hospital Administrator - staff member with an administrative role outside of the NICU leadership who is knowledgeable about the activities of the NICU NICU Manager - Nurse or physician with an administrative role in the NICU (e.g. medical director or nurse manager) H-HOPE Team member - staff member who is part of the H-HOPE Team NICU Staff Nurse - registered nurse who provides direct patient care and works a minimum of 50% in the NICU Exclusion Criteria We will not be limiting any participants based on sex/gender, or ethnic/racial identity. Differences due to race and gender will be accounted for during data analysis. We will be limiting enrollment to English or Spanish speaking parents due to the limited availability of valid measures for data collection in languages other than English and Spanish. However, we anticipate that we will still be able to recruit an ethnically diverse group of parents because of the ethnic composition of the parents at the sites and our prior experience.

Exclusion criteria for the infant:

* major brain injuries (e.g. cystic PVL)
* current sepsis
* intubated for mechanical ventilation at time of enrollment
* surgical necrotizing enterocolitis
* Ward of the State

Exclusion criteria for the parent:

* positive drug screen for illegal substances
* planning to surrender custody of the infant or legal custody remove
* primary parent does not have legal guardianship of the infant
* Mental health diagnosis such as Psychosis, Bipolar Disease Exclusion Criteria Hospital Personnel
* None

Exclusion Criteria for NICU Staff Nurses:

* less than 50% effort.
* does not provide direct patient care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1882 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Aim 1 Outcome Measure: Implementation Success (Percent Change in Sustainability throughout implementation) | Every 2 months from Executing through 6 months after supported implementation ends
  Change in % of instances of H-HOPE being offered
Aim 1 Outcome Measure: Implementation Success (Change in Reach throughout implementation) | Every 2 months from Executing through 6 months after supported implementation ends
  % of eligible parent-infant units receiving H-HOPE
Aim 1 Outcome Measure: Implementation Success (Degree of Implementation) | Every 2 months from Executing through 6 months after supported implementation ends
  In-Hospital:
  Infant: Mean number of ATVV interventions received per eligible day (Range 0-2)
  Transition to home:
  Parents: # received participatory guidance sessions (2 pre-discharge and 2 screen time visits at 2-3 days and 7-15 days post-discharge; Range: 0-3) Infant: Mean number of ATVV interventions received by per eligible day since discharge (Range 0-2; provided and reported by parent)
Aim 2 Outcome Measure: Effectiveness-(Change in Infant Head Circumference) | From birth to discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant)
  Infant Primary: Infant Head Circumference, measured in centimeters.
Aim 2 Outcome Measure: Effectiveness (Change in Infant Weight) | From birth to discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant)
  Infant Primary: Weight, measured in kilograms
Aim 2 Outcome Measure: Effectiveness (Change in Infant Length) | From birth to discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant)
  Infant Primary: Length, measured in centimeters
Aim 2 Outcome Measure: Effectiveness (Change in number of Acute Care Visits) | At 6 weeks post discharge
  Number of acute care visits (clinic or emergency department visit or re-hospitalization)

SECONDARY OUTCOMES:
Aim 2 Outcome Measure: Cost | From infant enrollment through infant discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant)
  Mean hospitalization cost/day (direct costs) from entry into H-HOPE through discharge, adjusted by adding the cost per H-HOPE infant to implement H-HOPE (training, coordinating, time to deliver H-HOPE and to arrange screen time visits)
Aim 3 Outcome Measure: CFIR influences (Number of facilitators and barriers to implementation) | From the completion of the first site's Sustaining Phase through Final Analysis of all site data, estimated to be 39 months.
  Aim 3 uses mixed methods analyses to integrate data collected for this aim regarding influences (facilitators or barriers) in each of the 5 CFIR domains with data from Aim 1 (implementation success) and Aim 2 (effectiveness for the primary infant outcomes).

OTHER OUTCOMES:
Aim 2 Exploratory Outcome Measure: # Parent NICU visits/days of hospitalization | At discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant)
  # Parent NICU visits/days of hospitalization (each parent)
Aim 2 Exploratory Outcome Measure: Parental Stress (Anxiety) | At discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant) and 6 weeks corrected Age
  PROMIS SF v1.0 - Anxiety7a
Aim 2 Exploratory Outcome Measure: Parental Stress (Depression) | At discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant) and 6 weeks corrected Age
  PROMIS SF v1.0 - Depression 8b
Aim 2 Exploratory Outcome Measure: Parental Stress (Child Health Worry Scale) | At discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant) and 6 weeks corrected Age
  Child Health Worry Scale. The scale values are 1=not worried; 2=somewhat worried; 3=moderately worried; 4=very worried; 5=extremely worried
Aim 2 Exploratory Outcome Measure: Confidence in Care | At discharge (an average of 31- 48 weeks PMA (Post Menstrual Age) of infant) and 6 weeks corrected Age
  (KPCS) Karitane Parenting Confidence Scale. The following choices are available to select for each of the scale's questions: No, hardly ever (0 points) , No, not very often (1 point), Yes, some of the time (2 points), Yes, most of the time (3 points). The points are added up and a total score is calculated. Parents with a total score of 39 or less may be experiencing low levels of parenting confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary White-Traut, PhD,RN,FAAN, Principal Investigator — Department of Nursing Research and Evidence-Based Practice Children's Wisconsin
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Advocate Aurora Health, Park Ridge, Illinois
  - Duke Univesity, Durham, North Carolina
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] White-Traut R, Brandon D, Kavanaugh K, Gralton K, Pan W, Myers ER, Andrews B, Msall M, Norr KF. Protocol for implementation of an evidence based parentally administered intervention for preterm infants. BMC Pediatr. 2021 Mar 24;21(1):142. doi: 10.1186/s12887-021-02596-1. PMID 33761902
- See also: Complete List of Published Work in MyBibliography for Rosemary White-Traut — https://www.ncbi.nlm.nih.gov/sites/myncbi/1zuy2pmUXmu5a/bibliography/48083153/public/?sort=date&direction=ascending